CLINICAL TRIAL: NCT04305015
Title: Postoperative Benefits of Intraoperative NOL Titration - Pilot
Brief Title: Postoperative Benefits of Intraoperative Nociception Level (NOL) Titration - Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medasense Biometrics Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLI-20-01
Record Dates: First submitted 2020-03-09; First posted 2020-03-12 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Nociceptive Pain
Keywords: NOL; Nociception
MeSH Terms: conditions — Nociceptive Pain

STUDY DESIGN:
Intervention Model Description: NOL-Guided analgesia vs. Routine Management
Who Masked: Participant, Outcomes Assessor
Masking Description: Anesthesia clinicians cannot be blinded since they will need to titrate opioid administration to NOL. However, all postoperative care and evaluations will be fully blinded to randomization, thus preventing measurement bias
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Routine opioid management (Active Comparator): Clinicians will be blinded to NOL monitoring and use clinical judgement to determine how much fentanyl should be given, and when
  Interventions: Other: Routine opioid management
- NOL-guided opioid administration (Experimental): Clinicians will titrate fentanyl to keep NOL under 25 - always using good clinical judgement for individual patients
  Interventions: Device: NOL Guided Analgesia

INTERVENTIONS:
Device: NOL Guided Analgesia — NOL values exceeding 25 will typically be treated with boluses of fentanyl 50 µg at roughly 5-minute intervals. The target will be maintained until surgery ends
  Other Names: Physiological Monitoring Device: PMD-200 system
  Arms: NOL-guided opioid administration
Other: Routine opioid management — Clinical judgement will be according to their standard practice and may include interpretation of blood pressure, heart rate, diaphoresis, tearing, and pupil size. Boluses of fentanyl 50 µg can be given per clinical judgement
  Arms: Routine opioid management

SUMMARY:
Previous work has shown that NOL (Medasense, Ramat Gan, Israel) accurately quantifies nociception during general anesthesia. Presumably, titrating opioids to NOL will therefore provide individual guidance so that patients will be given about the right amount. Patient given the right amount will presumably awaken quickly when anesthesia is done, and have good initial pain control in the post anesthesia care unit (PACU). To the extent that NOL titration facilitates optimal opioid dosing, patients are likely to have better PACU experiences - which would be an important outcome that clinicians and regulators are likely to take seriously.

ELIGIBILITY:
Inclusion Criteria:

1. Adults having major non-cardiac surgery expected to last ≥2 hours;
2. American Society of Anesthesiologists physical status 1-3;
3. Age 21-85 years old;
4. Planned endotracheal intubation

Exclusion Criteria:

1. Planned neuraxial or regional block;
2. Local anesthetic infiltration at surgical field;
3. Clinician preference for an opioid other than, or in addition to, fentanyl;
4. Non-sinus heart rhythm;
5. Neurologic condition that, in the opinion of the investigators, may preclude accurate assessment of postoperative pain and nausea;
6. Lack of English language fluency;
7. Routine user of psychoactive drugs other than opioids;
8. Contraindication to sevoflurane, fentanyl, morphine, or ondansetron.
9. Intracranial surgery
10. BMI > 40

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
PACU pain score | 60 minutes during recovery
  Average pain scores (0-10 verbal response scale) at 10-minute intervals during the initial 60 minutes of recovery are more often between 1 and 3 or significantly lower with NOL-guided fentanyl than with routine care

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No